CLINICAL TRIAL: NCT03628183
Title: Tolerance of Infants Fed a Hydrolysate Formula Manufactured With a New Processing Method
Brief Title: Tolerance of Infants Fed a Hydrolysate Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AL30
Record Dates: First submitted 2018-07-13; First posted 2018-08-14 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Gastrointestinal Tolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrolysate Infant Formula 1 (Active Comparator): Ready to feed infant formula in can
  Interventions: Other: Hydrolysate Infant Formula 1
- Hydrolysate Infant Formula 2 (Experimental): Ready to feed infant formula in bottle
  Interventions: Other: Hydrolysate Infant Formula 2

INTERVENTIONS:
Other: Hydrolysate Infant Formula 1 — Feed ad lib
  Arms: Hydrolysate Infant Formula 1
Other: Hydrolysate Infant Formula 2 — Feed ad lib
  Arms: Hydrolysate Infant Formula 2

SUMMARY:
This is a prospective, randomized, multicenter study to assess the tolerance of infant formulas.

ELIGIBILITY:
Inclusion Criteria:

* Subject is judged to be in good health
* Singleton from a full-term birth
* Birth weight was > or = to 2490 g
* Between 0 and 14 days of age at enrollment
* Parent(s) confirm their intention to feed their infant the assigned study product as the sole source of nutrition for the duration of the study
* Parent(s) confirm their intention not to administer vitamin or mineral supplements, solid foods or juices to their infant from enrollment through the duration of the study
* Subject's parent(s) has voluntarily signed and dated an Informed Consent Form (ICF)

Exclusion Criteria:

* An adverse maternal, fetal or subject medical history that is thought by the investigator to have potential for effects on tolerance, growth, and/or development.
* Subject is taking and plans to continue medications, home remedies, herbal preparations or rehydration fluids that might affect gastrointestinal (GI) tolerance
* Subject participates in another study that has not been approved as a concomitant study
* Subject has an allergy or intolerance to any ingredient in the study product
* Subject has been treated with antibiotics within 2 weeks prior to enrollment

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2018-11-23 (Actual)

PRIMARY OUTCOMES:
Stool Characteristics | Study Day 1 - Study Day 21
  Parent completed diary

SECONDARY OUTCOMES:
Formula Intake | Study Day 1 - Study Day 21
  Parent completed diary
Weight | Study Day 1 - Study Day 21
  Scale
Length | Study Day 1 - Study Day 21
  Length board

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Allgeier, MS, RD, LD, Study Chair — Abbott Nutrition
Locations (5):
- United States (5):
  - Watching Over Mothers and Babies, Tucson, Arizona
  - Springs Medical Research, Owensboro, Kentucky
  - The Cleveland Pediatric Research Center, LLC, Cleveland, Ohio
  - Institute of Clinical Research, LLC, Mentor, Ohio
  - Midsouth Center for Clinical Research, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided